CLINICAL TRIAL: NCT04380324
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Subcutaneous Dose of NKTR-358 in Healthy Volunteers
Brief Title: A Study of NKTR-358 (LY3471851) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17237; J1P-MC-KFAA (Other: Eli Lilly and Company); 16-358-01 (Other: Nektar Therapeutics)
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3471851 (Experimental): Healthy participants in each cohort will receive single subcutaneous (SC) doses of LY3471851.
  Interventions: Drug: LY3471851
- Placebo (Placebo Comparator): Healthy participants in each cohort will receive the placebo comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — LY3471851 drug product is a sterile liquid for SC injection that may be diluted with sterile 0.9% sodium chloride solution for injection (USP) prior to administration.
  Other Names: NKTR-358
  Arms: LY3471851
Drug: Placebo — The placebo dosing solution is 0.9% sodium chloride for injection (USP).
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of a study drug known as LY3471851 in healthy participants. The study will last about 50 days for each participant.

DETAILED DESCRIPTION:
LY3471851 is a potential first-in-class therapeutic that may address an underlying immune system imbalance in people with many autoimmune conditions. It targets the interleukin (IL-2) receptor complex in the body in order to stimulate proliferation of inhibitory immune cells known as regulatory T cells. By activating these cells, LY3471851 may act to bring the immune system back into balance.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males and females, as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.0 to 32.0 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Previous or current autoimmune disease/disorder
* Current active bacterial, viral, or fungal infection
* Administration of an inactivated vaccine within two weeks of study drug administration or live attenuated vaccine within 90 days of dosing .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Day 50
  Number of Participants with One or More SAEs Considered by the Investigator to be Related to Study Drug Administration

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3471851 | Predose on Day 1 through Day 50
  PK: Cmax of LY3471851
PK: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf]) of LY3471851 | Predose on Day 1 through Day 50
  PK: (AUC[0-inf]) of LY3471851
Pharmacodynamics (PD): Mean Change from Baseline in Regulatory T cells (Tregs) | Predose on Day 1 through Day 50
  PD: Mean change from baseline in Tregs
PD: Change from Baseline in Treg Activation Markers | Predose on Day 1 through Day 50
  PD: Treg activation markers include: Cytokine levels, conventional CD4+ and CD8+ Tcells, and natural killer (NK) cells

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No